CLINICAL TRIAL: NCT07351214
Title: THE EFFECT OF A MOTİVATİONAL İNTERVİEWİNG-BASED MİNDFULNESS İNTERVENTİON ON WEİGHT CONTROL AFTER BARİATRİC SURGERY: A RANDOMİZED CONTROLLED TRİAL.
Brief Title: THE EFFECT OF MOTİVATİONAL INTERVİEWİNG-BASED MİNDFULNESS INTERVENTION ON WEİGHT MANAGEMENT AFTER WEİGT LOSS,7SLİMMİNG SURGERY: A RANDOMİZED CONTROLLED TRIAL.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu Ateş (Other)
Responsible Party: Sponsor-Investigator, Duygu Ateş, LECTURER, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KA25/84
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Patients Who Gain Weight or Stop Losing Weight After barıatrıc Surgery; Absence of Cognitive or Psychiatric Illness; Not Having Previously Received Cognitive Awareness Training; Not Having Undergone Revision Surgery
Keywords: Obesity; Bariatric Surgery; Motivational Interviewing; Mindfulness
MeSH Terms: conditions — Mental Disorders; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): a mindfulness initiative based on motivational interviewing: Motivational interviewing over the phone three times, Mindfulness practices are face to face once a week for 8 weeks
  Interventions: Behavioral: A MİNDFULNESS İNİTİATİVE BASED ON MOTİVATİONAL İNTERVİEWİNG
- Control Group (No Intervention): standard training in an obesity clinic: In an obesity clinic, standard follow-up training is provided once a month by a dietitian, psychologist, nurse, and physiotherapist.

INTERVENTIONS:
Behavioral: A MİNDFULNESS İNİTİATİVE BASED ON MOTİVATİONAL İNTERVİEWİNG — Awareness initiatives were conducted face-to-face with 31 patients once a week for 8 weeks.
  Other Names: Awareness initiatives were conducted face-to-face with 31 patients once a week for 8 weeks.
  Arms: Intervention Group

SUMMARY:
Obesity is one of the most critical health problems in developed and developing countries, recognized as a chronic disease that adversely affects both individual and societal health. The World Health Organization (WHO) and other health authorities classify obesity based on Body Mass Index (BMI). Individuals with a BMI above 30 are categorized as obese, while those with a BMI above 40 are considered severely obese. Global statistics show a rapid increase in obesity prevalence, predicting that the number of obese individuals will reach 1.53 billion by 2035. In Turkey, the rate of women with high BMI has risen to 76%, and obesity prevalence has surpassed 30%.

Obesity is caused by unhealthy dietary habits, physical inactivity, genetic predisposition, and environmental factors, leading to serious health problems such as diabetes, hypertension, and cardiovascular diseases. Treatment methods include diet, exercise, medication, behavioral therapies, and surgical interventions. However, post-surgery patients are at risk of regaining lost weight if they fail to regulate their eating behaviors.

In recent years, motivational interviewing and mindfulness-based interventions have come to the forefront in obesity treatment. Motivational interviewing is an evidence-based technique that supports behavioral change by enhancing an individual's intrinsic motivation. Mindfulness-based approaches have proven effective in emotional regulation, stress management, and improving eating behaviors. Research has shown that these methods help post-bariatric surgery patients adjust their eating habits, maintain weight control, and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Literacy,
* Being between 18-65 years old,
* Regaining 5% or more of the minimum weight achieved at least 6 months after the surgery.

Exclusion Criteria:

* Having a diagnosed cognitive or psychiatric illness that would make it difficult for them to understand and adapt to the training content
* Having previously received cognitive awareness training
* Having undergone revision surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in weight loss maintenance awareness | Baseline and at 8 weeks after the intervention
  Awareness related to weight loss maintenance will be assessed using a validated awareness questionnaire administered by a trained researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will not share individual patient data as I believe it would be an ethical violation for the patients.